CLINICAL TRIAL: NCT05602038
Title: Comparative Study on the Effect of Quadratus Lumborum Block Versus Intrathecal Morphine on the Incidence of Chronic Pain Post Caesarean Section in a University Hospital of Middle-income Country; A Randomized Control Study
Brief Title: Comparative Study on the Effect of Quadratus Lumborum Block Versus Intrathecal Morphine on the Incidence of Chronic Pain Post Caesarean Section in a University Hospital of Middle-income Country
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2022ANET1-3
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Chronic Post Cesarean Pain

STUDY DESIGN:
Intervention Model Description: randomized control study
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients will be randomly allocated to the procedure through closed envelopes and so syringes and medication will be prepared and labelled by anesthetist other than the anesthetist giving the block
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group Q (Active Comparator): QLB group will receive 30 ml 0.125% bupivacaine (Sunnypivacaine by Sunny Pharmaceuticals) for each side
  Interventions: Procedure: Quadratus laborum block; Drug: intrathecal bupivacaine
- Group M (Active Comparator): Intrathecal morphine 100mcg will be added to bupivacaine 0.5% 15mg and fentanyl 20 µg
  Interventions: Drug: Intrathecal morphine; Drug: intrathecal bupivacaine
- Group QM (Active Comparator): Intrathecal morphine 100mcg will be added to bupivacaine 0.5% 15mg and fentanyl 20 µg combined by QLB of 30 ml 0.125%bupivacain
  Interventions: Procedure: Quadratus laborum block; Drug: Intrathecal morphine; Drug: intrathecal bupivacaine
- Group C (Placebo Comparator): Control group with intrathecal bupivacaine 0.5% 15mg and fentanyl 20 µg.
  Interventions: Drug: intrathecal bupivacaine

INTERVENTIONS:
Procedure: Quadratus laborum block — quadratus lumborum block will be performed using ultrasound machine (Sonosite Portable Ultrasound System, SonoSite, Bothell, Washington, USA). A 5-8 MHZ curved probe will be used with the patient positioned on the lateral side
  Arms: Group Q; Group QM
Drug: Intrathecal morphine — Intrathecal morphine 100mcg will be added to bupivacaine 0.5% 15mg and fentanyl 20 µg
  Arms: Group M; Group QM
Drug: intrathecal bupivacaine — intrathecal bupivacaine 0.5% 15mg and fentanyl

SUMMARY:
The aim of this study is to compare the incidence of CPSCP in patients receiving QLB quadratus lumborum block and ITM versus control as a primary outcome and associated risk factors that might predispose patients to develop CPSCP.

DETAILED DESCRIPTION:
The aim of this study is to compare the incidence of chronic post cesarean pain in patients receiving quadratus laborum block and and intrathecal morphine versus control as a primary

Study design:

Patients will be randomly allocated to the procedure through closed envelopes and so syringes and medication will be prepared and labelled by anesthetist other than the anesthetist giving the block Patients will be randomly allocated to the procedure through closed envelopes and so syringes and medication will be prepared and labelled by anesthetist other than the anesthetist giving the block Data will be collected regarding the demographic data, gestational stage, parity and number of previous cesarean section, previous abdominal surgeries, and narcotic consumption.

Postoperative pain day 1 and day2 will be followed by anesthetist who is blinded to the applied technique used. Follow up for the subsequent period of observation (2,4and 6 months) will be done by the department secretary who will contact the patients by phone to ask them if there is any "concern" after the operation. If the patient refers to a pain at the surgical site that has been lasting for the past three months a call will be conducted by the anesthetist and a referral schedule will be appointed to the pain clinic consultant for further evaluation

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the operating theatre for elective caesarean section

Exclusion Criteria:

* lack of informed consent
* Allergy to drugs used during the study
* Depression and epilepsy that required antidepressants or anticonvulsants
* known coagulopathy as a contraindication for spinal anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Post operative cesarean section pain
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Six months
  As zero is no pain and 10 is the maximum pain that can be felt

SECONDARY OUTCOMES:
narcotic consumption | 48 hours
  narcotic consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Menoufia, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No